CLINICAL TRIAL: NCT01853605
Title: NATRELLE® 410 Full and Moderate Height/Projection Breast Implant Continued Access Post-Approval Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was discontinued following product approval.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 410CA-002
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Results first posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-07

CONDITIONS: Breast Augmentation; Breast Reconstruction; Breast Implant Revision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Augmentation (Experimental): Women undergoing breast augmentation.
  Interventions: Device: Anatomically shaped silicone gel-filled breast implants
- Reconstruction (Experimental): Women undergoing breast reconstruction.
  Interventions: Device: Anatomically shaped silicone gel-filled breast implants
- Revision-Augmentation (Experimental): Women undergoing revision of previous breast augmentation.
  Interventions: Device: Anatomically shaped silicone gel-filled breast implants
- Revision-Reconstruction (Experimental): Women undergoing revision of previous breast reconstruction.
  Interventions: Device: Anatomically shaped silicone gel-filled breast implants

INTERVENTIONS:
Device: Anatomically shaped silicone gel-filled breast implants — Surgical implant
  Other Names: NATRELLE® 410 Highly Cohesive Anatomically Shaped Silicone-Filled Breast Implants (Styles 410 FM, FF, MM, or MF)

SUMMARY:
Post-approval study of the safety and effectiveness of NATRELLE® 410 Highly Cohesive Anatomically Shaped Silicone-Filled Breast Implants (Styles 410 FM, FF, MM, or MF) for breast augmentation, reconstruction, or revision

ELIGIBILITY:
Inclusion Criteria:

For entry in this study, subjects must have been enrolled in the 410 CA Clinical Study or 410 CARE Clinical Study under the inclusion criteria listed below and received NATRELLE® 410 Highly Cohesive Anatomically Shaped Silicone-Filled Breast Implants Styles 410 FM, FF, MM, or MF in 1 (for unilateral breast reconstruction or revision) or both breasts.

* Female, age 18 or older
* Present with one or more of the following conditions:
* Primary breast augmentation (i.e., no previous breast implant surgery) indicated for subject dissatisfaction, with size or shape of breast (e.g., mammary hypoplasia), asymmetry, ptosis, or aplasia
* Primary breast reconstruction (i.e., no previous breast implant surgery other than implantation of tissue expanders or contralateral augmentation for asymmetry) indicated, in the affected breast, for mastectomy for cancer, prophylactic mastectomy, or breast trauma (resulting in mastectomy) and for the unaffected breast, contralateral asymmetry (may be performed on the date of the mastectomy or the date when permanent implants are placed in the reconstructed breast)
* Breast implant revision surgery (i.e., removal and replacement of breast implants) indicated for previous augmentation or reconstruction with silicone-filled or saline-filled breast implants
* Has adequate tissue available to cover implants
* Willing to undergo MRI at the specified follow-up visit for subjects at MRI designated sites and be eligible for MRI (e.g., no implanted metal or metal devices, no history of severe claustrophobia)

Exclusion Criteria:

For entry in this study, subjects must have been enrolled in the 410 CA Clinical Study or 410 CARE Clinical Study and met the exclusion criteria listed below but not received any NATRELLE® 410 Highly Cohesive Anatomically Shaped Silicone-Filled 410 X- or L-Style Breast Implants

* Does not have advanced fibrocystic disease considered to be premalignant without accompanying subcutaneous mastectomy
* Does not have existing carcinoma of the breast, without mastectomy
* Does not have abscess or infection in the body at the time of enrollment
* Is not pregnant or nursing
* Does not have any disease, including uncontrolled diabetes (e.g., HbA1c > 8%), that is clinically known to impact wound healing ability
* Does not show tissue characteristics that are clinically incompatible with mammaplasty, such as tissue damage resulting from radiation, inadequate tissue, compromised vascularity, or ulceration
* Does not have or is under treatment for any condition that may constitute an unwarranted surgical risk (e.g., unstable cardiac or pulmonary problems)
* Does not show psychological characteristics that may be incompatible with the surgical procedure and the prosthesis, such as inappropriate attitude or motivation (e.g., body dysmorphic disorder)
* Is not willing to undergo further surgery for revision, if medically required

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3811 (Actual)
Dates: Start 2003-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan Medical
Locations (1):
- Eugene, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was discontinued following product approval.
Period: Overall Study
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Started | 1939 | 693 | 751 | 428
Completed | 1939 | 693 | 751 | 428
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction | Total
Number analyzed (Participants) | 1939 | 693 | 751 | 428 | 3811
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.0 (8.65) | 46.2 (9.96) | 49.8 (10.03) | 53.5 (9.11) | 42.5 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1939 | 693 | 751 | 428 | 3811
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Subject Satisfaction With Breast Implants on a 5-Point Scale
Description: Subject satisfaction with each breast implant is assessed on the following 5-point scale: (Definitely Satisfied, Somewhat Satisfied, Neither Satisfied nor Dissatisfied, Somewhat Dissatisfied, and Definitely Dissatisfied). Satisfaction is reported for subject's assessing satisfaction as definitely satisfied and somewhat satisfied. The worst response is used if the subject reports different responses for the left and right breasts.
Time Frame: 5 years
Population: Evaluable population: all enrolled subjects implanted with the NATRELLE 410 original style implants, who completed the 5 year follow-up visit, and had data at the time point.
Measure: Number; unit: Subjects
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Number analyzed (Participants) | 1929 | 688 | 740 | 419
Subjects
  Definitely Satisfied | 1772 | 559 | 542 | 295
  Somewhat Satisfied | 119 | 87 | 145 | 89

2. Primary Outcome: Investigator Satisfaction With Breast Implants on a 5-Point Scale
Description: Investigator satisfaction with each breast implant is assessed on the following 5-point scale: (Definitely Satisfied, Somewhat Satisfied, Neither Satisfied nor Dissatisfied, Somewhat Dissatisfied, and Definitely Dissatisfied). Satisfaction is reported for Investigator's assessing satisfaction as definitely satisfied and somewhat satisfied. The worst response is used if the Investigator reports different responses for the left and right breasts.
Time Frame: 5 years
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Number analyzed (Participants) | 1922 | 689 | 745 | 418
Subjects
  Definitely Satisfied | 1798 | 560 | 564 | 310
  Somewhat Satisfied | 97 | 83 | 141 | 83

3. Primary Outcome: Local Complications
Description: Local complications are the cumulative complications occurring in at least 5% of subjects in 1 or more cohorts over the duration of the study. The Kaplan-Meier risk rate is presented.
Time Frame: 5 years
Population: Evaluable population: all enrolled subjects implanted with the NATRELLE 410 original style implants who completed the 5 year follow-up visit.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Number analyzed (Participants) | 1939 | 693 | 751 | 428
Percentage of Subjects
  Capsular Contracture | 3.27 [2.56 to 4.16] | 6.33 [4.74 to 8.45] | 6.48 [4.92 to 8.51] | 7.29 [5.19 to 10.21]
  Asymmetry | 0.83 [0.51 to 1.35] | 0.87 [0.39 to 1.93] | 5.94 [4.46 to 7.90] | 3.32 [1.98 to 5.54]

ADVERSE EVENTS:
Description: Adverse event (AE) data experienced by ≥5% of subjects are recorded as an outcome measure.
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Serious Adverse Events (participants affected / at risk) | 0/1939 | 0/693 | 0/751 | 0/428
Other Adverse Events (participants affected / at risk) | 0/1939 | 0/693 | 0/751 | 0/428

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.